CLINICAL TRIAL: NCT02062411
Title: A Randomized Controlled Study of Cognitive Behavioral Therapy for Adults With Attention Deficit Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Sixth Hospital (Other)
Responsible Party: Principal Investigator, Qiujin Qian, PhD, Peking University Sixth Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2013-9-23-3
Record Dates: First submitted 2014-02-12; First posted 2014-02-13 (Estimated); Last update posted 2016-04-29 (Estimated); Status verified 2016-04

CONDITIONS: Attention Deficit Disorder
Keywords: attention deficit disorder (ADHD); cognitive behavioral therapy (CBT); adult
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- CBT with booster sessions (Experimental): Participants will receive 12 cognitive-behavioral therapy sessions weekly and 3 booster sessions monthly following our protocol.
  Interventions: Behavioral: CBT with booster sessions
- CBT only (Active Comparator): Participants will only receive 12 cognitive-behavioral therapy sessions weekly.
  Interventions: Behavioral: CBT only
- waiting (No Intervention): Participations will not be treated with CBT and keep waiting for 12 weeks for comparison.

INTERVENTIONS:
Behavioral: CBT only — Participants will learn 12 sessions including educational information about ADHD and skills in organization and plan, reducing distractibility, and adaptive thinking.
  Other Names: Mastering Your Adult ADHD manual (Safren, et al., 2005)
  Arms: CBT only
Behavioral: CBT with booster sessions — Participants are provided with the same CBT programme and additional 3 booster sessions which summarize and extend the 3 main topics of the CBT programme in order to improve the skills practice ability.
  Arms: CBT with booster sessions

SUMMARY:
The purpose of this study is to determine whether cognitive behavioral therapy (CBT) is effective in the treatment of attention deficit and emotional, executive function and social function dysregulation due to attention deficit disorder (ADHD).

DETAILED DESCRIPTION:
Participations will be randomly assigned to 3 groups which are CBT with booster sessions group, CBT only group and waiting group.With the comparison of first tow groups we will explore the effect of booster sessions, and the last two groups the effect of CBT programme.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients from Peking University Sixth Hospital
* Diagnosis of adult ADHD based on Diagnostic and statistical manual of mental disorders, Fourth Edition (DSM-IV)
* Stable on medications for adult ADHD for at least 2 months

Exclusion Criteria:

* Severe major depression, clinically significant panic disorder, bipolar disorder, organic mental disorders, psychotic disorders, or pervasive developmental disorders
* Intelligence Quotient (IQ) less than 90
* Suicide risk
* Unstable physical condition
* Prior participation in cognitive behavioral therapy for ADHD or other psychological therapy

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 108 (Actual)
Dates: Start 2013-10; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Change in ADHD Rating Scale | Baseline, at the end of week 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, and 11 in treatment, 12 weeks (post), 24 weeks (FU6), 36 weeks (FU9), and 48 weeks (FU12)
  ADHD symptom severity as measured by the ADHD rating scale (DuPaul, et al., 1998) a scale that ranges from 0-54 with 0 indicating lower severity.

SECONDARY OUTCOMES:
Change in Conners Adult ADHD Rating Scale Self-report Screening Version (CAARS-S:SV) | Baseline, at the end of week 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, and 11 in treatment, 12 weeks (post), 24 weeks (FU6), 36 weeks (FU9), and 48 weeks (FU12)
  The CAARS-S:SV is a self-reported scale measures the ADHD symptom severity including 30 items rating from 0 to 3.
Change in Self-Rating Anxiety Scale (SAS) | Baseline, at the end of week 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, and 11 in treatment, 12 weeks (post), 24 weeks (FU6), 36 weeks (FU9), and 48 weeks (FU12)
  The Self-Rating Anxiety Scale (SAS) with 20 items measures the level of anxiety.
Change in Self-rating depression scale (SDS) | Baseline, at the end of week 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, and 11 in treatment, 12 weeks (post), 24 weeks (FU6), 36 weeks (FU9), and 48 weeks (FU12)
  The Self-rating depression scale (SDS) is used to measure the level of depression.
Change in Behavior Rating Inventory of Executive Function-Adult Version (BRIEF-A) | Baseline, 12 weeks (post), 24 weeks (FU6), and 48 weeks (FU12)
  The BRIEF-A measures the impairment level of executive function in ADHD adults.
Change in Cambridge Neuropsychological Test Automatic Battery (CANTAB) | Baseline, 12 weeks (post), 24 weeks (FU6), and 48 weeks (FU12)
  The CANTAB is a computerized neuropsychological test measuring the cognitive and executive function.
Change in Barratt impulsiveness scale (BIS) | Baseline, 12 weeks (post), 24 weeks (FU6), and 48 weeks (FU12)
  The Barratt impulsiveness scale including 30 items is used to measure impulsiveness.
Change in self-esteem scale (SES) | Baseline, 12 weeks (post), 24 weeks (FU6), and 48 weeks (FU12)
  The self-esteem scale measures the level of self-esteem.
Change in World Health Organization Quality of Life-Brief Version (WHOQOL-BREF) | Baseline, 12 weeks (post), 24 weeks (FU6), and 48 weeks (FU12)
  The WHOQOL-BREF is the short version of World Health Organization Quality of Life scale and includes 26 items measuring the level of life quality.
Change in Brain Oxygenation Level Dependent (BOLD) Signal | Baseline, 12 weeks (post)
  The level of BOLD activity during working memory task after CBT is compared with baseline level to explore the potential effects of CBT on brain.

CONTACTS AND LOCATIONS:
Overall Officials: Qiujin Qian, PhD, Study Director — Peking University Sixth Hospital
Locations (1):
- Peking University Sixth Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Huang F, Qian Q, Wang Y. Cognitive behavioral therapy for adults with attention-deficit hyperactivity disorder: study protocol for a randomized controlled trial. Trials. 2015 Apr 14;16:161. doi: 10.1186/s13063-015-0686-1. PMID 25873090